CLINICAL TRIAL: NCT00619411
Title: An Open Clinical Trial of Interpersonal Psychotherapy for Depressed Adolescence and Parents
Brief Title: Interpersonal Psychotherapy for Depressed Adolescents and Parents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5549
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Major Depression; Dysthymic Disorder; Adjustment Disorders; Depressive Disorder Not Otherwise Specified
Keywords: Major Depression; Dysthymic Disorder; Adjustment Disorder; With Depressed Mood; Depressive; Disorder Not; Otherwise; Specified; Adolescent; Psychotherapy
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder; Adjustment Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental)
  Interventions: Behavioral: Interpersonal Therapy for Depressed Adolescents & Parents

INTERVENTIONS:
Behavioral: Interpersonal Therapy for Depressed Adolescents & Parents — 15 weekly psychotherapy sessions

SUMMARY:
The purpose of this study is to examine the feasibility and acceptability of an adaptation of Interpersonal Psychotherapy for Depressed Adolescents (IPT-A) that includes greater and more structured involvement of the parents in the treatment.

DETAILED DESCRIPTION:
Adolescent depression is a significant public health problem, and it increases the risk of poor psychosocial outcomes in adolescence and adulthood. Interpersonal Psychotherapy for Depressed Adolescents (IPT-A) has been found to be an effective treatment for reducing adolescents' depressive symptoms and improving their global and social functioning. The purpose of the current study is to examine the feasibility and acceptability of IPT-A when it is delivered with greater and more structured involvement of the parents in the treatment.

Participants will receive 15 weeks of Interpersonal Psychotherapy for Depressed Adolescents and Parents (IPT-AP). Eight the therapy sessions are conducted with the adolescent individually, two are with the parent(s) individually, and five are conducted with the adolescent and parent(s) together. At the end of the 15 weeks, participants who have demonstrated at least a 50% reduction in depressive symptoms will participate in three booster sessions delivered on a monthly basis. All participants will be assessed at baseline, week 5, week 10, week 15 (post-treatment), and 3 months post-treatment to measure depressive symptoms, global and social functioning, and attitudes toward treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for major depression, dysthymic disorder, depressive disorder not otherwise specified, or adjustment disorder with depressed mood
* Score between 10 and 28 on the HRSD
* Score of 65 or less on the C-GAS
* English-speaking adolescent
* Parental or legal guardian consent to participate

Exclusion Criteria:

* Actively suicidal
* Score greater than 28 on the HRSD
* Mentally retarded
* Meets diagnostic criteria for current substance abuse, schizophrenia, bipolar disorder, psychosis, conduct disorder, or eating disorder
* Currently in active treatment for depression
* Taking antidepressant medication at the time of baseline assessment
* Medical illness likely to complicate or interfere with treatment
* Victim of ongoing or previously undisclosed child abuse
* Parent psychiatrically hospitalized within the past 3 months

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2007-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Clinical Global Improvement (CGI), Hamilton Rating Scale for Depression (HRSD), Center for Epidemiological Studies - Depression Scale (CES-D) | baseline, week 5, 10, 15

SECONDARY OUTCOMES:
Global Assessment Scale for Children (C-GAS), Social Adjustment Scale - Self-report (SAS-SR), Conflict Behavior Questionnaire (CBQ-20), Observational assessment of parent-adolescent communication | baseline, week 5, 10, 15

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Gunlicks-Stoessel, Ph.D., Principal Investigator — University of Minnesota